CLINICAL TRIAL: NCT05335135
Title: Linking Novel Diagnostics With Data-Driven Clinical Decision Support in the Emergency Department
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Stocastic, LLC (Industry)
Collaborators: University of Kansas (Other); Beckman Coulter, Inc. (Industry); Truman Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 21-STOC-101
Record Dates: First submitted 2022-02-22; First posted 2022-04-19 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-03

CONDITIONS: Inpatient Hospitalization, Intensive Care Unit Admission, Inpatient Mortality, Sepsis and Septic Shock
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Pre-Implementation: Usual care will be provided during all ED patient encounters.
  Interventions: Other: Usual Care
- Post-Implementation: TriageGo-MDW CDS will be made available during all ED patient encounters at two points in the ED care continuum: (1) shortly after arrival during initial ED triage (First Triage) and (2) after initial laboratory results have been populated within the EHR. General illness severity estimates will be provided to nurses at ED triage in the form of recommended triage acuity scores (CDS for First Triage). General illness severity estimates along with estimated risk for specific outcomes including sepsis and septic shock will be presented to clinicians after laboratory results have populated (CDS for Early Assessment). TriageGO-MDW risk estimates will be generated by machine learning algorithms using routinely available clinical data as predictor inputs. Nurses and clinicians will receive risk estimates within existing EHR workflows, along with brief and rapidly interpretable explanations of the logic driving each risk estimate.
  Interventions: Other: TriageGO-MDW Clinical Decision Support

INTERVENTIONS:
Other: TriageGO-MDW Clinical Decision Support — TriageGO-MDW is non-device clinical decision support that provides patient-level clinical risk estimates based on clinical data derived from the electronic health record
  Groups: Post-Implementation
Other: Usual Care — Clinical care without decision support provided by TriageGo-MDW
  Groups: Pre-Implementation

SUMMARY:
The primary objective of this study is to validate the use of an electronic clinical decision support (CDS) tool, TriageGO with Monocyte Distribution Width (TriageGO-MDW), in the emergency department (ED). TriageGO-MDW is non-device CDS designed to support emergency clinicians (nurses, physicians and advanced practice providers) in performing risk-based assessment and prioritization of patients during their ED visit. This study will follow an effectiveness-implementation hybrid design via the following three aims (phases), to be executed sequentially:

(Aim 1) Validate the TriageGO-MDW algorithm locally using retrospective data at ED study sites.

(Aim 2) Deploy TriageGO-MDW integrated with the electronic medical record (EMR) and perform user assessment.

(Aim 3) Evaluate TriageGO-MDW in steady state with respect to clinical, process, and perceived utility outcomes.

ELIGIBILITY:
Inclusion Criteria: Adult patients receiving care at a study site ED

Exclusion Criteria: None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All emergency department visits by adult patients during the study period will be included in our analysis.
Sampling Method: Non-Probability Sample
Enrollment: 300000 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Critical Care | baseline (pre-intervention)
  Admission to an intensive care unit within 24 hours of ED disposition; Prediction performance of machine learning algorithms that underly TriageGO-MDW for this outcome will be measured
Critical Care | during post-implementation steady state (approximately 3 months after intervention)
  Admission to an intensive care unit within 24 hours of ED disposition; Prediction performance of machine learning algorithms that underly TriageGO-MDW for this outcome will be measured
In-Hospital Mortality | baseline (pre-intervention)
  Death during index hospital encounter; Prediction performance of machine learning algorithms that underly TriageGO-MDW for this outcome will be measured
In-Hospital Mortality | during post-implementation steady state (approximately 3 months after intervention)
  Death during index hospital encounter; Prediction performance of machine learning algorithms that underly TriageGO-MDW for this outcome will be measured
Emergent Surgery | baseline (pre-intervention)
  procedure in the operating room within 12 hours of ED arrival; Prediction performance of machine learning algorithms that underly TriageGO-MDW for this outcome will be measured
Emergent Surgery | during post-implementation steady state (approximately 3 months after intervention)
  procedure in the operating room within 12 hours of ED arrival; Prediction performance of machine learning algorithms that underly TriageGO-MDW for this outcome will be measured
Sepsis | baseline (pre-intervention)
  Prediction performance of machine learning algorithms that underlie TriageGO-MDW for this outcome will be measured
Sepsis | during post-implementation steady state (approximately 3 months after intervention)
  Prediction performance of machine learning algorithms that underlie TriageGO-MDW for this outcome will be measured
Septic Shock | baseline (pre-intervention)
  Meeting septic shock criteria within 24 hours of ED arrival; Prediction performance of machine learning algorithms that underly TriageGO-MDW for this outcome will be measured
Septic Shock | during post-implementation steady state (approximately 3 months after intervention)
  Meeting septic shock criteria within 24 hours of ED arrival; Prediction performance of machine learning algorithms that underly TriageGO-MDW for this outcome will be measured
Viral Infection | baseline (pre-intervention)
  Testing positive for influenza or Covid-19 (SARS-CoV-2) infection within 24 hours of ED arrival; Prediction performance of machine learning algorithms that underly TriageGO-MDW for this outcome will be measured
Viral Infection | during post-implementation steady state (approximately 3 months after intervention)
  Testing positive for influenza or Covid-19 (SARS-CoV-2) infection within 24 hours of ED arrival; Prediction performance of machine learning algorithms that underly TriageGO-MDW for this outcome will be measured

OTHER OUTCOMES:
Critical care triage capture rate | baseline (pre-intervention)
  Proportion of patients with critical care admission, emergency surgery or in-hospital mortality identified as high acuity at ED triage
Critical care triage capture rate | during post-implementation steady state (approximately 3 months after intervention)
  Proportion of patients with critical care admission, emergency surgery or in-hospital mortality identified as high acuity at ED triage
Hospital admission triage capture rate | baseline (pre-intervention)
  Proportion of patients requiring hospital admission identified as moderate or high acuity at ED triage
Hospital admission triage capture rate | during post-implementation steady state (approximately 3 months after intervention)
  Proportion of patients requiring hospital admission identified as moderate or high acuity at ED triage
ED patient flow metrics | baseline (pre-intervention)
  Intervals between major ED care events, including arrival to disposition, arrival to treatment space, arrival to treatment provider, arrival to intensive care unit transfer, arrival to ED departure will be measured
ED patient flow metrics | during post-implementation steady state (approximately 3 months after intervention)
  Intervals between major ED care events, including arrival to disposition, arrival to treatment space, arrival to treatment provider, arrival to intensive care unit transfer, arrival to ED departure will be measured
Sepsis care quality metrics | baseline (pre-intervention)
  Standard sepsis care quality metrics including time to diagnosis and treatment and rates of compliance with the Centers for Medicare and Medicaid Services (CMS) Sepsis-1 (SEP-1) Core Measure and its components will be measured
Sepsis care quality metrics | during post-implementation steady state (approximately 3 months after intervention)
  Standard sepsis care quality metrics including time to diagnosis and treatment and rates of compliance with the Centers for Medicare and Medicaid Services (CMS) Sepsis-1 (SEP-1) Core Measure and its components will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Scott Levin, PhD, Principal Investigator — Stocastic, LLC; Jeremiah Hinson, PhD/MD, Principal Investigator — Stocastic, LLC; Nima Sarani, MD, Principal Investigator — University of Kansas; Kevin O'Rourke, MD, Principal Investigator — Truman Medical Center
Locations (2):
- United States (2):
  - Kansas University Medical Center, Kansas City, Kansas
  - University Health Truman Medical Center, Kansas City, Missouri

REFERENCES:
- [Background] Levin S, Toerper M, Hamrock E, Hinson JS, Barnes S, Gardner H, Dugas A, Linton B, Kirsch T, Kelen G. Machine-Learning-Based Electronic Triage More Accurately Differentiates Patients With Respect to Clinical Outcomes Compared With the Emergency Severity Index. Ann Emerg Med. 2018 May;71(5):565-574.e2. doi: 10.1016/j.annemergmed.2017.08.005. Epub 2017 Sep 6. PMID 28888332
- [Background] Dugas AF, Kirsch TD, Toerper M, Korley F, Yenokyan G, France D, Hager D, Levin S. An Electronic Emergency Triage System to Improve Patient Distribution by Critical Outcomes. J Emerg Med. 2016 Jun;50(6):910-8. doi: 10.1016/j.jemermed.2016.02.026. Epub 2016 Apr 25. PMID 27133736
- [Background] Crouser ED, Parrillo JE, Seymour C, Angus DC, Bicking K, Tejidor L, Magari R, Careaga D, Williams J, Closser DR, Samoszuk M, Herren L, Robart E, Chaves F. Improved Early Detection of Sepsis in the ED With a Novel Monocyte Distribution Width Biomarker. Chest. 2017 Sep;152(3):518-526. doi: 10.1016/j.chest.2017.05.039. Epub 2017 Jun 15. PMID 28625579